CLINICAL TRIAL: NCT03054649
Title: A Prospective, Multicenter Study to Evaluate the Safety and Performance of the Exchangeable ClarVista HARMONI Modular Toric Intraocular Lens System for the Treatment of Pre-Existing Corneal Astigmatism and Aphakia Following Cataract Surgery
Brief Title: ClarVista HARMONI Toric Trial With Intraoperative Exchange
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ClarVista Medical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-00002
Record Dates: First submitted 2017-02-12; First posted 2017-02-15 (Actual); Results first posted 2020-06-22 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Cataract; Corneal Astigmatism; Aphakia
Keywords: cataract; intraoperative exchange; intraocular lens; astigmatism; toric
MeSH Terms: conditions — Cataract; Astigmatism; Aphakia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Cohort 1 (Experimental): Study eye: Primary implantation of HMIOL system with toric optic and no intraoperative optic exchange
  Interventions: Device: HARMONI® Modular Intraocular Lens System
- Cohort 2 (Experimental): Fellow eye: Primary implantation of HMIOL system with monofocal optic, followed by intraoperative optic exchange (toric or non-toric optic)
  Interventions: Device: HARMONI® Modular Intraocular Lens System; Procedure: Intraoperative optic exchange

INTERVENTIONS:
Device: HARMONI® Modular Intraocular Lens System — Two-component system consisting of a base and a separate optic that allows for an intraoperative exchange of the optic only without direct manipulation of the capsular bag
  Other Names: HMIOL
Procedure: Intraoperative optic exchange — Removal of one optic and replacement with another during cataract surgery for the purpose of improving refractive outcomes
  Other Names: IOE
  Arms: Cohort 2

SUMMARY:
The purpose of this study was to demonstrate the safety and effectiveness of the HARMONI® Modular Intraocular Lens System with a toric optic in subjects with pre-existing corneal astigmatism in need of cataract surgery.

DETAILED DESCRIPTION:
Subjects were implanted with the HARMONI® Modular Intraocular Lens System (HMIOL). The eye with the higher corneal astigmatism (study eye) was assigned to Cohort 1 and received the HARMONI® Modular Intraocular Lens System with a toric optic. The fellow eye was assigned to Cohort 2 and received the HARMONI® Modular Intraocular Lens System with a non-toric optic during primary implantation, which was replaced with the appropriate optic power (toric or non-toric) during an intraoperative exchange (IOE) procedure. A total of 7 study visits were planned, including a preoperative visit, operative visits for each eye, and 4 follow-up visits at 1 day, 1 week, 1 month, and 3 months postoperative. The total duration of participation for each subject was up to 6 months, which included a Day -90 to Day -0 preoperative period.

Alcon Research, LLC, acquired ClarVista Medical in 2017. This study was designed and conducted by ClarVista Medical, Inc. The study results were collected, analyzed, and provided by ClarVista Medical, Inc. to Alcon Research, LLC.

ELIGIBILITY:
Key Inclusion Criteria

* Willing and able to return for scheduled treatment and follow-up examinations for up to 6 month study duration.
* Planned removal of visually significant bilateral cataracts.
* Pre-existing corneal astigmatism in at least 1 eye.
* Willing to discontinue contact lens wear for the duration of the study.
* Best Corrected Visual Acuity (BCVA) projected to be 0.2 logarithm Minimum Angle of Resolution (logMAR) or lower.
* Visual symptoms related to cataracts.

Key Exclusion Criteria

* History of any intraocular or corneal surgery in either eye (including refractive).
* Pregnant or lactating.
* History of any clinically significant retinal pathology or ocular diagnosis in either eye that could alter or limit final postoperative visual prognosis.
* History of any ocular condition which could affect the stability of the intraocular lens (IOL) in either eye.
* Uncontrolled glaucoma in either eye (per Investigator judgement).
* Severe dry eye that, in the opinion of the investigator, would impair the ability to obtain reliable study measurements

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-06-28 (Actual); Primary Completion 2017-07-18 (Actual); Study Completion 2017-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Clinical Trial Lead, CDMA Surgical, Study Director — Alcon Research, LLC
Locations (2):
- ClarVista Investigative Site, Tijuana, Estado de Baja California, Mexico
- ClarVista Investigative Site, Makati, Manila, Philippines

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 1 site located in the Philippines and 1 site located in Mexico. Of the 44 subjects signing an informed consent, 12 failed to meet inclusion/exclusion criteria and 5 were withdrawn prior to implantation when the intraocular lens power was not available due to inventory restrictions.
Pre-assignment Details: This reporting group includes all implanted subjects/eyes. Note: One eye in Cohort 2 attempted implantation but was discontinued due to capsular instability (preferred term: Ciliary zonular dehiscence), which was reported as an intraoperative SAE.
Units Other Than Participants: eyes
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 27; 27 eyes | 27; 26 eyes
Completed | 27; 27 eyes | 27; 26 eyes
Not Completed | 0; 0 eyes | 0; 0 eyes

BASELINE CHARACTERISTICS:
Population: All implanted subjects
Groups:
- HMIOL: Implantation with HMIOL system
Arm/Group | HMIOL
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.4 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 25
  Black | 0
  Caucasian | 0
  Other | 2

OUTCOME MEASURES:

1. Primary Outcome: Mean Manifest Refraction Cylinder (MRCYL) for Eyes Implanted With HMTIOL
Description: A manifest refraction (manual vision test) was conducted using letter charts and a phoropter. Manifest refraction cylinder is the amount of added correction needed to compensate for any astigmatism that may be present. MRCYL was measured in diopters and reported as a negative number, with a less negative number indicating a lesser amount of added correction. No formal statistical hypothesis testing was planned.
Time Frame: Month 1 postoperative, Month 3 postoperative
Population: Per Protocol: All eyes with successful implantation of the HMTIOL and no major protocol deviations.
Measure: Mean (Standard Deviation); unit: diopter
Units Other Than Participants: eyes
Groups:
- Cohort 2: Fellow eye: Primary implantation of HMIOL system with monofocal optic, followed by intraoperative optic exchange (toric optic)
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 27 | 15
Number analyzed (eyes) | 27 | 15
diopter
  Month 1 postoperative | -0.54 (0.32) | -0.75 (0.31)
  Month 3 postoperative | -0.58 (0.42) | -0.72 (0.45)

2. Primary Outcome: Mean Manifest Refraction Cylinder (MRCYL) Prediction Error (PE) for Eyes Implanted With HMTIOL
Description: A manifest refraction (manual vision test) was conducted using letter charts and a phoropter. Manifest refraction cylinder is the amount of power needed to correct any astigmatism that may be present. MRCYL was measured in diopters and reported as a negative number. MRCYL PE was calculated as postoperative MRCYL adjusted to 6 meters minus MRCYL target residual refractive error (TRRE), with a lower absolute value indicating a more accurate cylinder power calculation. No formal statistical hypothesis testing was planned.
Time Frame: Month 1 postoperative, Month 3 postoperative
Population: Per Protocol: All eyes with successful implantation of the HMTIOL and no major protocol deviations.
Measure: Mean (Standard Deviation); unit: diopter
Units Other Than Participants: eyes
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 27 | 15
Number analyzed (eyes) | 27 | 15
diopter
  Month 1 postoperative | -0.30 (0.28) | -0.53 (0.36)
  Month 3 postoperative | -0.33 (0.33) | -0.44 (0.37)

3. Primary Outcome: Mean Reduction in Cylinder Power for Eyes Implanted With HMTIOL
Description: A manifest refraction (manual vision test) was conducted using letter charts and a phoropter. Manifest refraction cylinder is the amount of power needed to correct any astigmatism that may be present. MRCYL was measured in diopters and reported as a negative number. Cylinder power reduction was calculated as the absolute preoperative magnitude of corneal cylinder (K) minus the absolute postoperative magnitude of MRCYL at the corneal plane. No formal statistical hypothesis testing was planned.
Time Frame: Baseline (Day 0 preoperative), Month 3 postoperative
Population: Per Protocol: All eyes with successful implantation of the HMTIOL and no major protocol deviations.
Measure: Mean (Standard Deviation); unit: diopter
Units Other Than Participants: eyes
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 27 | 15
Number analyzed (eyes) | 27 | 15
diopter | 0.79 (0.56) | 0.53 (0.39)

4. Primary Outcome: Mean Percent Reduction in Cylinder Power for Eyes Implanted With HMTIOL
Description: A manifest refraction (manual vision test) was conducted using letter charts and a phoropter. Manifest refraction cylinder is the amount of power needed to correct any astigmatism that may be present. MRCYL was measured in diopters and reported as a negative number. Cylinder power reduction was calculated as the absolute preoperative magnitude of corneal cylinder (K) minus the absolute postoperative magnitude of MRCYL at the corneal plane. Therefore, the cylindrical power percent reduction was the cylinder power reduction divided by the absolute value of preoperative magnitude of corneal cylinder (K) × 100. A higher number (greater percent reduction) indicates better astigmatism correction by the toric IOL. No formal statistical hypothesis testing was planned.
Time Frame: Baseline (Day 0 preoperative), Month 3 postoperative
Population: Per Protocol: All eyes with successful implantation of the HMTIOL and no major protocol deviations.
Measure: Mean (Standard Deviation); unit: percent reduction
Units Other Than Participants: eyes
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 27 | 15
Number analyzed (eyes) | 27 | 15
percent reduction | 54.9 (29.3) | 39.5 (34.2)

5. Primary Outcome: Mean Manifest Refraction Spherical Equivalent (MRSE) Prediction Error (PE)
Description: A manifest refraction (manual vision test) was conducted using letter charts and a phoropter. The manifest refraction spherical equivalent (MRSE) was calculated as follows: sphere + 1/2 cylinder, and measured in diopters (D). MRSE PE was calculated as postoperative MRSE adjusted to 6 meters minus MRSE target residual refractive error (TRRE). The lower the absolute number, the more accurate the IOL power calculation is. No formal statistical hypothesis testing was planned.
Time Frame: Month 3 postoperative
Population: Implanted Eye Set: All eyes with successful implantation during surgery, with data at visit
Measure: Mean (Standard Deviation); unit: diopter
Units Other Than Participants: eyes
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 27 | 26
Number analyzed (eyes) | 27 | 26
diopter | 0.03 (0.45) | -0.12 (0.43)

6. Primary Outcome: Mean Absolute Rotation of IOL Meridian
Description: IOL orientation was measured with slit-lamp photography. IOL rotation was defined as the difference between axis of IOL orientation on the day of surgery and the subsequent postoperative visit. IOL rotation was measured in degrees, with a lower number indicating less rotation. No formal statistical hypothesis testing was planned.
Time Frame: Baseline (Day 0 operative), Day 1 postoperative, Week 1 postoperative, Month 1 postoperative, Month 3 postoperative
Population: Implanted Eye Set: All eyes with successful implantation during surgery, with data at visit
Measure: Mean (Standard Deviation); unit: degrees
Units Other Than Participants: eyes
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 24 | 20
Number analyzed (eyes) | 24 | 20
degrees
  Rotation from operative to Day 1: number analyzed (eyes) | 22 | 20
  Rotation from operative to Day 1 | 1.8 (1.3) | 2.1 (1.4)
  Rotation from operative to Week 1: number analyzed (eyes) | 23 | 17
  Rotation from operative to Week 1 | 2.4 (1.4) | 1.6 (1.7)
  Rotation from operative to Month 1: number analyzed (eyes) | 24 | 18
  Rotation from operative to Month 1 | 3.1 (4.5) | 2.3 (1.5)
  Rotation from operative to Month 3: number analyzed (eyes) | 23 | 19
  Rotation from operative to Month 3 | 3.2 (4.6) | 2.2 (1.6)

7. Primary Outcome: Number of Eyes With Absolute Rotation of IOL Meridian by Visit - Cohort 1
Description: IOL orientation was measured with slit-lamp photography. IOL rotation was defined as the difference between axis of IOL orientation on the day of surgery and the subsequent postoperative visit. IOL rotation was measured in degrees and is reported categorically. No formal statistical hypothesis testing was planned.
Time Frame: Baseline (Day 0 operative), Day 1 postoperative, Week 1 postoperative, Month 1 postoperative, Month 3 postoperative
Population: Implanted Eye Set: All eyes with successful implantation during surgery, with data at visit
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Groups:
- Cohort 1 - Day 1 Postoperative; Cohort 1 - Week 1 Postoperative; Cohort 1 - Month 1 Postoperative; Cohort 1 - Month 3 Postoperative: Study eye: Primary implantation of HMIOL system with toric optic and no intraoperative optic exchange
Arm/Group | Cohort 1 - Day 1 Postoperative | Cohort 1 - Week 1 Postoperative | Cohort 1 - Month 1 Postoperative | Cohort 1 - Month 3 Postoperative
Number analyzed (Participants) | 22 | 23 | 24 | 23
Number analyzed (eyes) | 22 | 23 | 24 | 23
eyes
  Rotation from Operative ≤ 5 degrees | 22 | 23 | 23 | 22
  Rotation from Operative >5 degrees to ≤ 10 degrees | 0 | 0 | 0 | 0
  Rotation from Operative >10 degrees to ≤ 20 degree | 0 | 0 | 0 | 0
  Rotation from Operative > 20 degrees | 0 | 0 | 1 | 1

8. Primary Outcome: Number of Eyes With Absolute Rotation of IOL Meridian by Visit - Cohort 2
Description: as for outcome 7
Time Frame: Baseline (Day 0 operative), Day 1 postoperative, Week 1 postoperative, Month 1 postoperative, Month 3 postoperative
Population: Implanted Eye Set: All eyes with successful implantation during surgery, with data at visit
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Groups:
- Cohort 2 - Day 1 Postoperative; Cohort 2 - Week 1 Postoperative; Cohort 2 - Month 1 Postoperative; Cohort 2 - Month 3 Postoperative: Fellow eye: Primary implantation of HMIOL system with monofocal optic, followed by intraoperative optic exchange (toric or non-toric optic)
Arm/Group | Cohort 2 - Day 1 Postoperative | Cohort 2 - Week 1 Postoperative | Cohort 2 - Month 1 Postoperative | Cohort 2 - Month 3 Postoperative
Number analyzed (Participants) | 20 | 17 | 18 | 19
Number analyzed (eyes) | 20 | 17 | 18 | 19
eyes
  Rotation from Operative ≤ 5 degrees | 20 | 17 | 18 | 19
  Rotation from Operative >5 degrees to ≤ 10 degrees | 0 | 0 | 0 | 0
  Rotation from Operative >10 degrees to ≤ 20 degree | 0 | 0 | 0 | 0
  Rotation from Operative > 20 degrees | 0 | 0 | 0 | 0

9. Primary Outcome: Percentage of Eyes With Best Corrected Distance Visual Acuity (BCDVA) by Visit - Cohort 1
Description: Visual Acuity of the eye was tested while reading charts at 20-foot equivalent distance from the participant with the correction obtained from manifest refraction testing. BCDVA is reported categorically using the Snellen fraction, which compares the participant's result to the result expected from a 'normal' visual system. The numerator represents the distance between the participant and the chart, and the denominator represents the distance at which a person with 'normal' vision would be able to discern the same letter size. 20/20 is considered to be 'normal' vision, whereas visual acuity of 20/40 means the participant is able to read a certain size letter 20 feet away that a person with 'normal' vision would be able to read from 40 feet away. A larger denominator, therefore, indicates a lower visual acuity. No formal statistical hypothesis testing was planned.
Time Frame: Baseline (Day 0 operative), Week 1 postoperative, Month 1 postoperative, Month 3 postoperative
Population: Implanted Eye Set: All eyes with successful implantation during surgery, with data at visit
Measure: Number; unit: Percentage of eyes
Units Other Than Participants: eyes
Groups:
- Cohort 1 - Baseline (Day 0 Preoperative); Cohort 1 - Week 1 Postoperative; Cohort 1 - Month 1 Postoperative; Cohort 1 - Month 3 Postoperative: Study eye: Primary implantation of HMIOL system with toric optic and no intraoperative optic exchange
Arm/Group | Cohort 1 - Baseline (Day 0 Preoperative) | Cohort 1 - Week 1 Postoperative | Cohort 1 - Month 1 Postoperative | Cohort 1 - Month 3 Postoperative
Number analyzed (Participants) | 27 | 27 | 27 | 27
Number analyzed (eyes) | 27 | 27 | 27 | 27
Percentage of eyes
  20/20 Snellen or Better | 22.2 | 66.7 | 59.3 | 70.4
  20/25 Snellen or Better | 51.9 | 77.8 | 85.2 | 92.6
  20/32 Snellen or Better | 70.4 | 96.3 | 100.0 | 96.3
  20/40 Snellen or Better | 92.6 | 100.0 | 100.0 | 96.3
  Worse than 20/40 Snellen | 7.4 | 0.0 | 0.0 | 3.7

10. Primary Outcome: Percentage of Eyes With Best Corrected Distance Visual Acuity (BCDVA) by Visit - Cohort 2
Description: Visual Acuity of the eye was tested while reading charts at 20-foot equivalent distance from the participant with the correction obtained from manifest refraction testing. UCDVA is reported categorically using the Snellen fraction, which compares the participant's result to the result expected from a 'normal' visual system. The numerator represents the distance between the participant and the chart, and the denominator represents the distance at which a person with 'normal' vision would be able to discern the same letter size. 20/20 is considered to be 'normal' vision, whereas visual acuity of 20/40 means the participant is able to read a certain size letter 20 feet away that a person with 'normal' vision would be able to read from 40 feet away. A larger denominator, therefore, indicates a lower visual acuity. No formal statistical hypothesis testing was planned.
Time Frame: Baseline (Day 0 operative), Week 1 postoperative, Month 1 postoperative, Month 3 postoperative
Population: Implanted Eye Set: All eyes with successful implantation during surgery, with data at visit
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Groups:
- Cohort 2 - Baseline (Day 0 Preoperative); Cohort 2 - Week 1 Postoperative; Cohort 2 - Month 1 Postoperative; Cohort 2 - Month 3 Postoperative: Fellow eye: Primary implantation of HMIOL system with monofocal optic, followed by intraoperative optic exchange (toric or non-toric optic)
Arm/Group | Cohort 2 - Baseline (Day 0 Preoperative) | Cohort 2 - Week 1 Postoperative | Cohort 2 - Month 1 Postoperative | Cohort 2 - Month 3 Postoperative
Number analyzed (Participants) | 26 | 26 | 26 | 26
Number analyzed (eyes) | 26 | 26 | 26 | 26
percentage of eyes
  20/20 Snellen or Better | 23.1 | 76.9 | 73.1 | 76.9
  20/25 Snellen or Better | 57.7 | 84.6 | 88.5 | 92.3
  20/32 Snellen or Better | 76.9 | 96.2 | 92.3 | 100
  20/40 Snellen or Better | 88.5 | 96.2 | 100.0 | 100.0
  Worse than 20/40 Snellen | 11.5 | 3.8 | 0.0 | 0.0

11. Primary Outcome: Percentage of Eyes With Uncorrected Distance Visual Acuity (UCDVA) by Visit - Cohort 1
Description: Visual Acuity of the eye was tested while reading charts at 20-foot equivalent distance from the participant with an optical infinity adjustment of +0.25 diopter (D). The Snellen fraction compares the participant's result to the result expected from a 'normal' visual system. The numerator represents the distance between the participant and the chart, and the denominator represents the distance at which a person with 'normal' vision would be able to discern the same letter size. 20/20 is considered to be 'normal' vision, whereas visual acuity of 20/40 means the participant is able to read a certain size letter 20 feet away that a person with 'normal' vision would be able to read from 40 feet away. A larger denominator, therefore, indicates a lower visual acuity. No formal statistical hypothesis testing was planned.
Time Frame: Baseline (Day 0 operative), Day 1 postoperative, Week 1 postoperative, Month 1 postoperative, Month 3 postoperative
Population: Implanted Eye Set: All eyes with successful implantation during surgery, with data at visit
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Groups:
- Day 1 Postoperative; Cohort 1 - Week 1 Postoperative; Cohort 1 - Month 1 Postoperative; Cohort 1 - Month 3 Postoperative: Study eye: Primary implantation of HMIOL system with toric optic and no intraoperative optic exchange
Arm/Group | Cohort 1 - Baseline (Day 0 Preoperative) | Day 1 Postoperative | Cohort 1 - Week 1 Postoperative | Cohort 1 - Month 1 Postoperative | Cohort 1 - Month 3 Postoperative
Number analyzed (Participants) | 27 | 27 | 27 | 27 | 27
Number analyzed (eyes) | 27 | 27 | 27 | 27 | 27
percentage of eyes
  20/20 Snellen or Better | 3.7 | 48.1 | 44.4 | 40.7 | 40.7
  20/25 Snellen or Better | 14.8 | 55.6 | 59.3 | 74.1 | 70.4
  20/32 Snellen or Better | 14.8 | 77.8 | 88.9 | 92.6 | 92.6
  20/40 Snellen or Better | 40.7 | 96.3 | 100.0 | 96.3 | 96.3
  Worse than 20/40 Snellen | 59.3 | 3.7 | 0.0 | 3.7 | 3.7

12. Primary Outcome: Percentage of Eyes With Uncorrected Distance Visual Acuity (UCDVA) by Visit - Cohort 2
Description: as for outcome 11
Time Frame: Baseline (Day 0 operative), Day 1 postoperative, Week 1 postoperative, Month 1 postoperative, Month 3 postoperative
Population: Implanted Eye Set: All eyes with successful implantation during surgery, with data at visit
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Cohort 2 - Baseline (Day 0 Preoperative) | Cohort 2 - Day 1 Postoperative | Cohort 2 - Week 1 Postoperative | Cohort 2 - Month 1 Postoperative | Cohort 2 - Month 3 Postoperative
Number analyzed (Participants) | 26 | 26 | 26 | 26 | 26
Number analyzed (eyes) | 26 | 26 | 26 | 26 | 26
percentage of eyes
  20/20 Snellen or Better | 0.0 | 46.2 | 53.8 | 42.3 | 34.6
  20/25 Snellen or Better | 3.8 | 65.4 | 76.9 | 73.1 | 69.2
  20/32 Snellen or Better | 11.5 | 65.4 | 84.6 | 88.5 | 84.6
  20/40 Snellen or Better | 50.0 | 92.3 | 92.3 | 100.0 | 100.0
  Worse than 20/40 Snellen | 50.0 | 7.7 | 7.7 | 0.0 | 0.0

13. Primary Outcome: Number of Eyes With Preservation of BCDVA at Month 1 and Month 3
Description: Preservation of BCDVA was defined in terms of lines lost when reading the ETDRS chart at each visit compared to the prior best-achieved BCDVA. Loss of < 1 line included subjects with less than a 1 line loss, no change or improvement in BCDVA. No formal statistical hypothesis testing was planned.
Time Frame: Week 1 postoperative, Month 1 postoperative, Month 3 postoperative
Population: All implanted subjects/eyes
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Cohort 1 - Month 1 Postoperative | Cohort 1 - Month 3 Postoperative | Cohort 2 - Month 1 Postoperative | Cohort 2 - Month 3 Postoperative
Number analyzed (Participants) | 27 | 27 | 26 | 26
Number analyzed (eyes) | 27 | 27 | 26 | 26
eyes
  Loss < 1 line | 27 | 25 | 25 | 26
  Loss >= 1 lines | 0 | 2 | 1 | 0
  Loss >= 2 lines | 0 | 1 | 0 | 0
  Loss >= 3 lines | 0 | 0 | 0 | 0
  Loss >= 4 lines | 0 | 0 | 0 | 0

14. Primary Outcome: Number of Ocular Adverse Events Through Month 3
Description: Ocular adverse events were identified as outlined in ISO 11979-2014 Annex B. No formal statistical hypothesis testing was planned.
Time Frame: Up to Month 3 postoperative
Population: Safety Analysis Set: All subjects/eyes with attempted study lens implantation (successful or aborted).
Measure: Number; unit: adverse event
Units Other Than Participants: eyes
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 27 | 27
Number analyzed (eyes) | 27 | 27
adverse event
  Conjunctivitis viral | 1 | 0
  Cystoid macular oedema | 1 | 1
  Ciliary zonular dehiscence | 0 | 1
  Intraocular pressure increased | 0 | 1
  Iridocyclitis | 0 | 1

15. Primary Outcome: Number of Device Deficiencies Post Implantation
Description: A Device Deficiency (DD) was defined as a failure of the device to meet its performance specifications or expectations, or otherwise not perform as intended. This could include either a malfunction or damage to the device or any part thereof, regardless of the source of malfunction or damage, including user error, and regardless of the presence of injury (or lack thereof) to subject, user, or bystander. No formal statistical hypothesis testing was planned.
Time Frame: Up to Month 3 postoperative
Population: All implanted subjects/eyes
Measure: Number; unit: device deficiency
Units Other Than Participants: eyes
Groups:
- Cohort 1 - No Exchange: Study eye: Primary implantation of HMIOL system with toric optic and no intraoperative optic exchange
- Cohort 2 - Intraoperative Exchange: Fellow eye: Primary implantation of HMIOL system with monofocal optic, followed by intraoperative optic exchange (toric or non-toric optic)
Arm/Group | Cohort 1 - No Exchange | Cohort 2 - Intraoperative Exchange
Number analyzed (Participants) | 27 | 26
Number analyzed (eyes) | 27 | 26
device deficiency | 0 | 0

16. Primary Outcome: Number of Secondary Surgical Interventions, Other Than Intraroperative Optic Exchange and Rotational Adjustment of the Toric Optic in Cohort 2
Description: A secondary surgical intervention (SSI) was defined as a surgical procedure that occurred after primary implantation and was conducted for the purpose of resolving residual refractive error (RRE) and optimizing visual outcomes. No formal statistical hypothesis testing was planned.
Time Frame: Up to Month 3 postoperative
Population: All implanted subjects/eyes
Measure: Number; unit: Secondary surgical interventions
Units Other Than Participants: eyes
Arm/Group | Cohort 1 - No Exchange | Cohort 2 - Intraoperative Exchange
Number analyzed (Participants) | 27 | 27
Number analyzed (eyes) | 27 | 27
Secondary surgical interventions | 0 | 0

17. Primary Outcome: Percent Change in Endothelial Cell Count (ECC) at Month 3
Description: High quality images of the corneal endothelium (the single layer of cells on the inner surface of the cornea) were taken at the investigative site and sent to an independent central reading center for evaluation. A negative percent change value may indicate a decrease in the ability of the endothelium to maintain its primary function. No formal statistical hypothesis testing was planned.
Time Frame: Baseline (preoperative), Month 3 postoperative
Population: All implanted subjects/eyes
Measure: Mean (Standard Deviation); unit: percent change
Units Other Than Participants: eyes
Arm/Group | Cohort 1 - No Exchange | Cohort 2 - Intraoperative Exchange
Number analyzed (Participants) | 27 | 26
Number analyzed (eyes) | 27 | 26
percent change | -12.5 (10.1) | -9.0 (10.3)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from time of consent until study exit: Up to 6 months, including a Day -90 to Day -0 preoperative period and a 3-month postoperative period.
Description: An adverse event was defined as any untoward medical event that does not necessarily have a causal relationship to the study device or protocol. Conditions or diseases that were pre-existing and/or chronic but stable were not recorded as adverse events. Similarly, changes in a pre-existing and/or chronic condition or disease that were consistent with natural progression were not recorded as adverse events.
Arm/Group | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27 | 1/27
Other Adverse Events (participants affected / at risk) | 0/27 | 0/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=27) | Cohort 2 (N=27)
Eye complication associated with device (General disorders) | 0 (0) | 1 (1) — Implantation attempted but discontinued due to capsular instability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2016-12-01): https://cdn.clinicaltrials.gov/large-docs/49/NCT03054649/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-14): https://cdn.clinicaltrials.gov/large-docs/49/NCT03054649/SAP_001.pdf